CLINICAL TRIAL: NCT00751998
Title: A Clinical Registry to Assess Performance and Clinical Utility of the SpyGlass Direct Visualization System
Brief Title: Spy II Clinical Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7012
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Biliary Tract Diseases
Keywords: biliary; ERCP; cholangioscopy; pancreatic
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Arm 1: Test of SpyGlass device
  Interventions: Device: SpyGlass

INTERVENTIONS:
Device: SpyGlass — The SpyGlass Direct Visualization System is an integrated product platform that is designed to provide a direct intraluminal view of the biliary duct system and direct therapeutic devices.

SUMMARY:
A prospective, multi-center registry for subjects undergoing Endoscopic retrograde Cholangiopancreatography (ERCP) and cholangioscopy for known or suspected pancreaticobiliary disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age
* Willing and able to comply with the Registry procedures and provide written informed consent to participate in the Registry
* Indicated for ERCP or ERCP/cholangioscopy (with or without biopsy)

Exclusion Criteria:

* Subjects for whom endoscopic procedure are medically contraindicated
* Subjects for whom ERCP are medically contraindicated
* Subjects for whom medical condition warrants use of device outside of indication for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are undergoing ERCP or ERCP/cholangioscopy for known or suspected pancreaticobiliary disease.
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Peetermans, PhD, Study Director — Boston Scientific Corporation
Locations (15):
- United States (10):
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Indiana University Medical Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Erasme Hospital - Belgium, Brussels, Belgium
- Bispebjerg Hospital, Denmark, København NV, Denmark
- Hopital Edouard Herriot, Lyon, France
- Evangelisches Krankenhaus Dusseldorf, Düsseldorf, Germany
- Policlinico Agostino Gemelli, Roma, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 27, 2006 and April 4, 2008 a total of 297 subjects were enrolled.
Period: Overall Study
Arm/Group | Arm 1
Started | 297
Completed | 277
Not Completed | 20
Not completed — Lost to Follow-up | 7
Not completed — Death | 11
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 157
  >=65 years | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 145
Region of Enrollment [Number; unit: participants]
  France | 15
  United States | 224
  Belgium | 11
  Denmark | 10
  Germany | 26
  Italy | 11

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success as Defined by: 1. Ability to Visualize Stricture & Obtain Biopsy of Lesion Adequate for Histological Examination in Suspected Malignancy Cases or 2. Ability to Visualize Stone(s) & Successfully Initiate Stone Fragmentation & Removal.
Time Frame: During Procedure
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm 1
Number analyzed (Participants) | 297
percent | 89 [84 to 92]

ADVERSE EVENTS:
Time Frame: 2 Years, 5 Months, & 17 Days
Description: Adverse Events were collected from procedure through end of study for all subjects.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 81/297
Other Adverse Events (participants affected / at risk) | 0/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=297)
Stent Migration (Hepatobiliary disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Escherichia Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Bacterial Sepsis (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Heparin induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Septicemia (Infections and infestations) | 3 (3)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1) — from ovarian cancer
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — From Ovarian Cancer
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Bell's Palsy (Nervous system disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Worsening of Left C5-6 Radiculopathy (Nervous system disorders) | 1 (1)
Fever (Infections and infestations) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 15 (15)
End Stage Liver Disease (Hepatobiliary disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Carcinamatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1)
Perforation of Bile Duct (Hepatobiliary disorders) | 1 (1) — From ERCP guidewire.
Abdominal Pain (Gastrointestinal disorders) | 5 (7)
Elevated Liver Function Tests (Hepatobiliary disorders) | 2 (2)
Hepatitis C (Hepatobiliary disorders) | 1 (1)
Liver Transplant Rejection (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2) — Unknown Type
Progression of malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Abdominal Aortic Aneurysm Repair with Stent Graft (Vascular disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Bile Duct Resection due to Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abdominal Distress (Gastrointestinal disorders) | 1 (1)
Unknown Cardiovascular Event (Cardiac disorders) | 1 (1) — resulting in death
Obstruction of Bile Duct (Hepatobiliary disorders) | 5 (5)
Transient Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 2 (2)
Liver Abcess (Hepatobiliary disorders) | 4 (4)
Probable Ileus (Gastrointestinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Diagnosis of Cancer of the Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pericarditis and effusion (Cardiac disorders) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 1 (1)
Umbilical Hernia Repair (Musculoskeletal and connective tissue disorders) | 1 (1)
Duct of Luschka Biliary Leak with Extrahepatic Biliary Stricture (Hepatobiliary disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Biliary Stent Replacement (Hepatobiliary disorders) | 3 (3)
Esophageal Variceal Bleeding (Gastrointestinal disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Choledocal Cyst (Hepatobiliary disorders) | 1 (1)
Delayed Return of Bowel Function (Gastrointestinal disorders) | 1 (1)
Biloma with Possible Superinfection (Infections and infestations) | 1 (1)
Post ERCP Nausea (Injury, poisoning and procedural complications) | 1 (1)
Intra-abdominal Hemorrhage Post Planned Surgical Intervention (Gastrointestinal disorders) | 1 (1)
Probable Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Inflammatory Syndrome (Immune system disorders) | 4 (6)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Dysfunction of Pancreatic Stent (Hepatobiliary disorders) | 1 (1)
Hospitalization for EUS and Abdominal Ultrasound (Gastrointestinal disorders) | 1 (1)
Hospitalization to Repeat ERCP & Continue Bile Duct Investigation (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No